CLINICAL TRIAL: NCT03710330
Title: A Double-blind, Placebo-controlled, Randomized Clinical Trial Comparing a Standard 1gm and a Low Dose 0.5gm IV Tranexamic Acid for the Control of Blood Loss at Elective Cesarean Section
Brief Title: Tranexamic Acid for the Control of Blood Loss at Elective Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/276/7/18
Record Dates: First submitted 2018-10-13; First posted 2018-10-18 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Eligible participants were allocated to one of three groups after induction of general anesthesia and immediately prior to the operation and just before skin incision. Groups were labeled as follows:
  Group one (120) - 5 ml of distilled water in 20 ml of 5% dextrose
  Group two (120) - TA in the dose of I gm in 20 ml of 5% dextrose
  Group three(120) - TA in the dose of 0.5gm in 20 ml of 5% dextrose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal saline (Placebo Comparator): the patients receives 110 ml normal saline IV just before skin incision
  Interventions: Drug: normal saline
- 1gm tranexamic acid (Active Comparator): 1 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision
  Interventions: Drug: 1gm tranexamic acid
- 0.5 gm tranexamic acid (Active Comparator): 0.5 gm tranexamic acid (1 ampoule of Capron 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision
  Interventions: Drug: 0.5 gm tranexamic acid

INTERVENTIONS:
Drug: normal saline — 110 ml normal saline IV just before skin incision
  Other Names: placebo comparator
  Arms: normal saline
Drug: 1gm tranexamic acid — 1 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision
  Other Names: active comparator
  Arms: 1gm tranexamic acid
Drug: 0.5 gm tranexamic acid — 0.5 gm tranexamic acid (2 ampoules of Capron 500 mg /5 ml; Cairo, Egypt) intravenous just before skin incision
  Other Names: active comparator
  Arms: 0.5 gm tranexamic acid

SUMMARY:
The aim of the study is to determine, out of two doses (a standard and a low dose) compared to placebo, the optimal and minimal dose of an intravenously administered single bolus of tranexamic acid(TA) to reduce blood loss when administered during cesarean section(CS). Tranexamic acid is an antifibrinolytic agent, which causes a reversible and competitive blockade of the lysine binding sites on plasminogen molecules. It is a synthetic analog of the amino acid lysine and its action is to reduce blood loss. TA is widely in use in the field of obstetrics. Both antepartum and postpartum hemorrhage(PPH) is being treated by TA extensively. One study demonstrated for the first time that TA administered to women with overt PPH decreases blood loss and maternal morbidity. Prevention of PPH is another indication where TA has been used. Varied doses of TA ranging from 1 mg/kg to more than 100 mg/kg have been used in various surgeries. Even in studies involving CS, the doses used were either a bolus of 1 gm or 10 mg/kg intravenously.

The dose of 1 g or 10 mg/kg is commonly used prophylactically before CS, Because of the lack of data on lower doses and TA pharmacokinetics, a low 0.5-g dose should be tested.

DETAILED DESCRIPTION:
CS was carried out under subarachnoid block using 2-2.5 ml of 0.5% hyperbaric bupivacaine after an informed written consent. Blockade up to T4-T6 level was considered an adequate level of anesthesia. After delivery of the neonate, 20 unit of oxytocin in 500 ml normal saline will begive at the rate of 8 mU/min intravenously.

All consenting patients were recruited as a consecutive series to one of the three study groups of 120 patients each, based on block random allocation protocol. Neither the patient nor the investigator was aware of the group assignment. An anesthesiologist not related to the study prepared the drug for every patient.

Groups were labeled as follows:

Group one (120) - 5 ml of distilled water in 20 ml of 5% dextrose

Group two (120) - TA in the dose of I gm in 20 ml of 5% dextrose

Group three(120) - TA in the dose of 0.5gm in 20 ml of 5% dextrose.

The drug in all the groups was given intravenously over 20 min before skin incision.

Monitoring of the pulse rate, blood pressure, Pulse Oximetry (SpO2) and Electrocardiograph (ECG) was carried out every 2 min up to 10 min of starting the study drug; then every 5 min until the delivery of the baby and thereafter every 15 min until the end of the surgery. Blood loss was measured intra-operatively and postoperatively up to 24 h. All material such as sponges, mops, pads, and drapes were weighed with an electronic weighing scale before and at the end of surgery. A volume of blood in the suction bottle was considered only after the placental delivery, to exclude any amniotic fluid volume. The quantity of intra-operative blood loss (ml) = (weight of the abdominal swabs and drapes after CS - weight of materials prior to CS) + (the volume in the suction bottle after placental delivery in ml). Post-operative blood loss was measured by weighing and numbering the vaginal pads used by the patient after completion of CS 2 hourly up to 6 h and then 6 hourly up to 24 h.

Uterine contractility, placental separation, neonatal condition and any side effect caused by TA will be noted. Intramuscular methylergometrine would be used as a rescue uterotonic treatment when required. Post-operative hemoglobin, hematocrit, serum creatinine, and prothrombin time, values were recorded at 24 h. All the parturients were encouraged to start early leg exercises and ambulation in the post-operative period.

ELIGIBILITY:
Inclusion Criteria: all pregnant women scheduled for elective cesarean -

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease.
* patients had an allergy to tranexamic acid

  . -patients who had received platelet antiaggregant such as Aspirin in the week before surgery
* patient refusing to be a participant

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — all pregnant women scheduled for elective cesarean
Enrollment: 360 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  amount of blood loss during the operation

SECONDARY OUTCOMES:
postoperative blood loss | 6 hours post operative
  amount of blood loss 6 hours post operative
Number of participants need of uterotonic | 24 hours post operative
  Number of participants need of extra uterotonic
Number of participants need blood transfusion | 24 hours post operative
  Number of participants need of blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No